CLINICAL TRIAL: NCT00893802
Title: Influence of Periodontal Treatment in Pregnant Women Attending Antenatal Care at a Public Health Center in Adverse Pregnant Outcomes: a Controlled Clinical Trial
Brief Title: Influence of Periodontal Treatment During Pregnancy in Adverse Pregnant Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Adriana Campos Passanezi Sant'Ana, Discipline of Periodontics, School of Dentistry at Bauru-USP
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP102/2002/FOB; CEP 102/2002
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2009-05-06 (Estimated); Status verified 2009-05

CONDITIONS: Periodontal Disease
Keywords: periodontal disease; pregnancy; periodontal treatment
MeSH Terms: conditions — Periodontal Diseases | interventions — Tooth Exfoliation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Periodontal treatment (Experimental): Scaling and root planning
  Interventions: Other: Scaling and root planning
- Control (No Intervention)

INTERVENTIONS:
Other: Scaling and root planning — Intervention will consist of supra and subgingival scaling and root planning performed by a single trained periodontist using Gracey curettes (Hu-Friedy, Chicago, USA) without local or general anesthesia during the second trimester of gestation, followed by professional prophylaxis and oral hygiene instruction. Treatment will be performed only once during study.
  Arms: Periodontal treatment

SUMMARY:
The aim of this study is to evaluate the effects of treatment of periodontal disease during the second trimester of gestation in adverse pregnancy outcomes.

Pregnant patients during the 1st and 2nd trimesters at antenatal care in a Public Health Center will be divided into two groups: NIG- 'no intervention' or IG- 'intervention,' according to agreement in receive periodontal treatment during pregnancy. Treatment will be performed by a single periodontist consisting of scaling and root planning (SRP), professional prophylaxis (PROPH) and oral hygiene instruction (OHI). Patients at NIG will receive PROPH and OHI during pregnancy and will be referred for treatment after delivery. Periodontal evaluation will be performed by a single trained examiner, blinded to periodontal treatment, according to probing depth (PD), clinical attachment level (CAL), plaque index (PI) and sulcular bleeding index (SBI) at baseline and 35 gestational weeks-28 days post-partum. Primary adverse pregnancy outcomes to be addressed are: preterm birth (< 37 weeks), low birth weight (< 2.500 Kg), late abortion (14-24 weeks) or abortion (< 14 weeks). The results obtained will be statistically evaluated according to OR, unpaired t test and paired t test.

It is expected that periodontal treatment during the second trimester of gestation will result in decreased rates of adverse pregnancy outcomes.

DETAILED DESCRIPTION:
All patients entering the study at the 1st and 2nd trimesters will be invited to participate in an oral health program, including oral hygiene instruction, caries diagnosis and treatment, and evaluation and treatment of periodontal conditions during the second trimester. Those who refuse to receive periodontal treatment during pregnancy will constitute the 'no intervention' control group (NIG), while those who agree in receiving dental and periodontal treatment during the second trimester of gestation will constitute the 'intervention' group (IG).

Patients are going to be evaluated by a single calibrated periodontist blinded in relation to periodontal treatment, which will be performed by another periodontist. Treatment consists of scaling and root planning, professional prophylaxis and oral hygiene instruction. Obstetrical data, birth weight and gestation duration will be recorded after examination and recording by the responsible obstetrician and nursery staff.

ELIGIBILITY:
Inclusion Criteria:

* confirmed singleton gestations
* pregnancy of 9-24
* systemically healthy women
* age range: 16-39 years old

Exclusion Criteria:

* non confirmed pregnancy
* age inferior to 16 years or superior to 39 years
* multiple gestations
* smoking
* alcohol or drugs abuse
* history of congenital heart disease
* current use of corticosteroids or antibiotics
* presence of systemic conditions (eg: diabetes, hypertension, or genitor-urinary infections)

Ages: 16 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2001-08; Primary Completion 2002-08 (Actual); Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Primary outcome measures recorded are: preterm birth (PTB), defined as delivery < 37 weeks; low birth weight (LBW), defined as < 2.500Kg birth weight; preterm birth and low birth weight | Within 30 days after delivery

SECONDARY OUTCOMES:
Secondary outcome measures are: late abortion (14-24 gestational weeks); and abortion (< 14 gestational weeks) | Within 30 days after development

CONTACTS AND LOCATIONS:
Overall Officials: Adriana P Sant'Ana, DDS PhD, Study Director — Associate Professor - School of Dentistry at Bauru-USP; Marinele R Campos, DDS, Principal Investigator — Graduation student on Periodontics (Master level). School of Dentistry at Bauru - USP
Locations (1):
- Jardim Redentor I Public Health Center, Bauru, São Paulo, Brazil